CLINICAL TRIAL: NCT02231892
Title: Repetitive Transcranial Magnetic Stimulation Equipment Testing and Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 999914186; 14-DA-N186 (Other: NIDA)
Record Dates: First submitted 2014-09-03; First posted 2014-09-04 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2019-09-18

CONDITIONS: Healthy Volunteer
Keywords: Repetitive TMS (rTMS); Parameter Development; Cognitive Tasks; MRI (Magnetic Resonance Imaging)

STUDY DESIGN:
Intervention Model Description: Within-subject design with each subject completing up to 10 rTMS sessions.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Real TMS (Experimental): rTMS (frequency and intensity)
  Interventions: Device: TMS
- Sham TMS (Sham Comparator): Sham setting on coil
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — HAC coil (real rTMS or sham rTMS)

SUMMARY:
Background:

- Brain stimulation called repetitive transcranial magnetic stimulation (rTMS) may help people quit drugs. Researchers want to study how it works in healthy people first.

Objective:

- To learn how to use rTMS to stimulate a brain area and to see how it affects brain function and thinking.

Eligibility:

- Healthy, right-handed adults ages 18-55.

Design:

* Participants will be screened under another protocol.
* They will have 4-11 study visits.
* To start each visit, participants will have:
* Physical exam.
* Urine sample.
* Breath tests for alcohol and cigarette smoke.
* Questions about drug use and medications.
* Visit 1: participants will have:
* Single TMS pulses on the head to determine the right strength. They will wear earplugs and a cap. A wire coil will be placed on the head and an electrical current will go through it. Participants may perform simple muscle movements. They will repeat the procedures wearing another coil, in a helmet.
* A few TMS pulses to show how rTMS feels.
* A practice thinking task, maybe in a scanner that looks and sounds like a magnetic resonance imaging (MRI) scanner but does not take pictures. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. The participant will lie on a table that slides in and out of the cylinder.
* They may have a real MRI scan.
* Visits 2-11, participants will:
* Complete two questionnaires.
* Get varied rTMS stimulation. Their heart rate and blood pressure may be monitored.
* Have their vital signs checked.
* They may perform thinking tasks at a computer, in a mock scanner, or in an MRI scanner. They may just lie still in the MRI scanner.

DETAILED DESCRIPTION:
Objective: To establish an effective repetitive transcranial magnetic stimulation (rTMS) protocol for stimulating circuits relevant for addiction. Specifically, we will develop stimulation parameters and outcome measures for rTMS of the anterior cingulate cortex (ACC) with a specialized TMS coil: the HAC coil (Brainsway Ltd.). Various parameters of rTMS stimulation (frequency and intensity) will be varied, and the sensitivity of behavioral tasks and MRI measures to this stimulation will be determined. The objective of this protocol is therefore to allow for the development, assessment and refinement of rTMS parameters for stimulating ACC targets. In addition, outcome measures will be developed to capture the effects of this stimulation. Results from this development protocol will be applied to subsequent cognitive imaging protocols.

Study population: Up to 50 healthy, non-smoking adults will be tested in several conditions over up to two weeks. Subjects must fit exclusion/inclusion criteria for TMS and MRI. We expect 140 subjects to be enrolled to arrive at a number of 50 who complete the protocol.

Design: Within-subject design with each subject completing up to 10 rTMS sessions.

Outcome measures: In a first phase, the outcome measure will be the behavioral response on a task that relies on the ACC. In a second phase, outcome measures will be the effects on MR measures. These will include task-related blood oxygen level-dependent (BOLD) responses, as well as resting state BOLD functional magnetic resonance imaging (fMRI). Other MR measures, such as magnetic resonance spectroscopy (MRS) and arterial spin labeling (ASL), will also be explored as potential biomarkers.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must:

1. Be able to give valid informed consent
2. Be 18 55 years of age.

   1. Justification: Many neural processes change with age, and these changes could introduce unwanted variability in both behavioral and MRI signals. In addition, the risk of difficult-to-detect medical abnormalities such as silent cerebral infarcts increases with age.
   2. Screening tool: History. Government-issued forms of identification (e.g. driver s license, birth certificate) will be required when participant appears to be out of age range.
3. Be in good health.

   1. Justification: Many illnesses may alter neural functioning as well as fMRI signals.
   2. Screening tools: Medical Assessment, Medical History and Physical Examination. Medical assessments include: Vital Signs, EKG, oral HIV test, height/weight measurements, urinalysis and blood sample. Tests on the blood sample include complete blood count (CBC), complete metabolic profile, thyroid-stimulating hormone (TSH), erythrocyte sedimentation rate (ESR), Serologic Test For Syphilis (STS) and HIV (if needed to confirm a positive salivary test for HIV). The following individual laboratory results will independently disqualify individuals: Cholesterol >250 mg/dl, Hemoglobin < 10.5 g/dl, white blood cell count (WBC) < 2400/microl, liver function tests (LFTs) > 3x normal, Human chorionic gonadotropin (HCG) positive, Casual serum glucose > 200 mg/dl, Urine protein > 1+. The medically accountable investigator (MAI) will retain discretion to exclude at less extreme values, depending on the clinical presentation. (Serum glucose over 140 mg/dl will be followed up with a fasting serum glucose assessment. Those with fasting glucose below 100 mg/dl may be considered for the protocol. Others will be rejected and referred for work-up.) MAI will make the final judgment on any questionable lab results.
4. Right-handed.

   1. Justification: Using right-handed individuals will reduce variability in BOLD MRI data.
   2. Screening tool: Edinburgh Handedness Inventory.
5. Estimated intelligence quotient (IQ) greater than or equal to 85

   1. Justification: Subjects must be able to perform a cognitively challenging task to a high standard.
   2. Screening tool: Wechsler Abbreviated Scale of Intelligence.

EXCLUSION CRITERIA:

1. Personal history of stroke, brain lesions, previous neurosurgery, any personal history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than two days.

   Justification: Stroke or head trauma can lower the seizure threshold, and are therefore contra-indications for TMS. Fainting episodes or syncope of unknown cause could indicate an undiagnosed condition associated with seizures.

   Screening tool: TMS adult safety questionnaire, Medical History.
2. First-degree family history of any neurological disorder with a potentially hereditary basis, including migraines, epilepsy, or multiple sclerosis.

   1. Justification: Neurological disorders can lower the seizure threshold, and are therefore contra-indications for TMS. First-degree family history of certain neurological disorders with a hereditary component increases the risk of the subject having an undiagnosed condition that is associated with lowered seizure threshold.
   2. Screening tool: TMS adult safety screening, Medical History.
3. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head that precludes MRI scanning.

   1. Justification: Any metal around the head is a contraindication for both MRI and TMS, as both methods involve exposure to a relatively strong magnetic field.
   2. Screening tool: TMS adult safety screening, MRI safety screening, Medical History.
4. Noise-induced hearing loss or tinnitus.

   1. Justification: individuals with noise-induced hearing problems may be particularly vulnerable to the acoustic noise generated by TMS and MRI equipment.
   2. Screening tools: TMS adult safety screening.
5. Current use (any use in the past 4 weeks, chronic use within 6 past six months) of any investigational drug or of any medications with psychotropic, anti or pro-convulsive action.

   1. Justification: The use of certain medications or drugs can lower seizure threshold and is therefore contra-indicated for TMS.
   2. Screening tools: MRI safety screening questionnaire, Medical history, Medical Assessments: Urine toxicology analyzes for presence of a broad range of prescription and nonprescription drugs.
6. Lifetime history of major depressive disorder, schizophrenia, bipolar disorder, mania, or hypomania.

   1. Justification: The population of interest here is a healthy control population with no psychiatric disorders. In subjects with depression, bipolar disorder, mania or hypomania, there is a small chance that TMS can trigger (hypo)manic symptoms.
   2. Screening tools: Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID) Screen Patient Questionnaire. Potential diagnoses will be further evaluated by a counsellor.
7. Meet current Diagnostic and Statistical Manual (DSM) V criteria for moderate to severe substance use disorder (excluding nicotine), smoke daily, or urine toxicology positive for any illicit substance inconsistent with history given.

   1. Justification: The population of interest here is a healthy control population with no substance use disorder. Current use of illicit substances could impact on seizure threshold and is therefore contra-indicated for TMS.
   2. Screening tools: SCID Screen Patient Questionnaire. Potential diagnoses will be further evaluated by a counsellor, Drug Use Survey (DUS), Substance Use Disorder Evaluation, Medical Assessments: urine qualitative drug screen is performed for methadone, benzodiazepines, cocaine, amphetamine/methamphetamine, opiates, barbiturates, and tetrahydrocannabinol.
8. Have met DSM V criteria for moderate to severe substance use disorder (excluding nicotine, alcohol and cannabis) in the past, or have met DSM V criteria for moderate to severe substance use disorder for cannabis or alcohol in the past 5 years.

   1. Justification: the population of interest here is a healthy control population with no present or past substance use disorder.
   2. Screening tools: SCID Screen Patient Questionnaire. Potential diagnoses will be further evaluated by a counselor. Drug Use Survey (DUS), Substance Use Disorder Evaluation.
9. History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or any heart condition currently under medical care.

   1. Justifications: the risk of TMS for individuals with a heart condition is unknown.
   2. Screening tool: physical assessment (EKG), medical history.
10. Pregnant women or women with reproductive potential who are sexually active and not using an acceptable form of contraception.

    1. Justification: it is unknown whether TMS poses a risk to fetuses.
    2. Screening tool: Medical assessments (urine pregnancy test) at the beginning of each visit that involves TMS or MRI.
11. History of learning disability or current attention deficit hyperactivity disorder (ADHD)

    1. Justification: Subjects should be able to perform cognitive tasks to a high degree of accuracy, both in the MRI scanner and outside the scanner. Subjects with ADHD/LD may engage different neural circuitry even if they can perform the tasks.
    2. Screening tool: Wechsler Abbreviated Scale of Intelligence, Medical history, Adult ADHD Self-Report Scale.
12. Participation in an rTMS session less than two weeks ago.

    1. Justification: in order to limit exposure to TMS, we will not enroll subjects who have received TMS less than two weeks ago.
    2. Screening tool: TMS safety screening questionnaire.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2014-09-03; Primary Completion 2019-01-03 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Orientation occurred prior to starting repetitive transcranial magnetic stimulation (rTMS) days. Orientation consisted of single-pulse TMS (allowed participant to experience TMS and researcher to find motor hotspot) and habituation (allowed participant to habituate to varied TMS intensities). Many ppts withdrew or were excluded during orientation.
Groups:
- Low Frequency rTMS - Behavioral Phase: Participants in this arm received sham or active 1 hertz (Hz) rTMS at 100% and 110% of motor threshold during the behavioral phase.
- High Frequency rTMS - Behavioral Phase: Participants in this arm received sham or active 10 hertz (Hz) rTMS at 100% and 110% of motor threshold during the behavioral phase
- High Frequency rTMS - MRI Phase: Participants in this arm received sham or active 10 hertz (Hz) rTMS at 100% and 110% of motor threshold during the MRI phase of the study.
Period: Overall Study
Arm/Group | Low Frequency rTMS - Behavioral Phase | High Frequency rTMS - Behavioral Phase | High Frequency rTMS - MRI Phase
Started | 17 | 17 | 70
Sham (All participants were randomly assigned to sham, 100% MT, or 110% MT on each of 3 Study Days.) | 8 | 5 | 26
100% MT (All participants were randomly assigned to sham, 100% MT, or 110% MT on each of 3 Study Days.) | 7 | 6 | 25
110% MT (All participants were randomly assigned to sham, 100% MT, or 110% MT on each of 3 Study Days.) | 7 | 5 | 27
Completed | 6 | 5 (3 participants completed this phase and Hi Frequency MRI phase, but are only counted in Hi Freq MRI.) | 25 (3 participants completed this phase and Hi Frequency Beh phase, but are only counted in Hi Freq MRI.)
Not Completed | 11 | 12 | 45
Not completed — Lost to Follow-up | 1 | 0 | 3
Not completed — Withdrawal by Subject | 4 | 3 | 15
Not completed — Physician Decision | 0 | 2 | 4
Not completed — Motor activity when stimulating ante ACC | 4 | 7 | 12
Not completed — Participant motor threshold was >83% | 0 | 0 | 9
Not completed — Could not find motor threshold | 2 | 0 | 1
Not completed — Could not find reliable motor hotspot | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Frequency rTMS - Behavioral Phase: Participants in this arm received sham or active 1Hz rTMS at 100% and 110% of motor threshold during the behavioral phase
- High Frequency rTMS - Behavioral Phase: Participants in this arm received sham or active 10Hz rTMS at 100% and 110% of motor threshold during the behavioral phase
- High Frequency rTMS - MRI Phase: Participants in this arm received sham or active 10Hz rTMS at 100% and 110% of motor threshold during the MRI phase of the study.
- Total: Total of all reporting groups
Arm/Group | Low Frequency rTMS - Behavioral Phase | High Frequency rTMS - Behavioral Phase | High Frequency rTMS - MRI Phase | Total
Number analyzed (Participants) | 17 | 17 | 70 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 2 | 2
  Between 18 and 65 years | 17 | 17 | 68 | 102
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30.12 [21 to 48] | 28.55 [19 to 55] | 32.39 [18 to 55] | 31.27 [18 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 39 | 56
  Male | 9 | 8 | 31 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 6 | 10
  Not Hispanic or Latino | 15 | 15 | 64 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 8 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 14 | 12 | 36 | 62
  White | 2 | 3 | 25 | 30
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 70 | 104

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Outcome Measure
Description: Behavioral effects of INTENSITY (Sham/100%MT/110%MT) and demand for cognitive control, DEMAND (High/Medium/Low), were planned to be quantified via correct response time (RT) and trial accuracy using R Project for Statistical Computing (package afex, function mixed (Singmannet al, 2015)). RT data were planned to be submitted to a linear mixed model with a random intercept per subject and fixed effects of INTENSITY and DEMAND. Accuracy data were planned to be submitted to a generalized linear mixed model with a binomial distribution and logit link function with a random intercept per subject and fixed effects of INTENSITY and DEMAND.
  During the Behavioral phase of the study, this data was collected before TMS, immediately after TMS, and 1 hour after TMS. During the MRI phase of the study, this data was only collected before TMS and immediately after TMS.
Time Frame: 3x per session in Behavioral phase (before TMS, immediately after TMS, and 1 hour after TMS), and 2x per session in MRI Phase (before TMS and immediately after TMS).
Population: Data have not yet been analyzed due to personnel turnover. There are currently no resources to complete data analysis at this time. We have transferred data to a repository protocol for future analysis when resources for data analysis are available.
Arm/Group | Low Frequency rTMS - Behavioral Phase | High Frequency rTMS - Behavioral Phase | High Frequency rTMS - MRI Phase
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Imaging Outcome Measures
Description: These measures include resting state (seed-based functional connectivity), Arterial Spin labeling (ASL), and MRI Spectroscopy (MRS).
  1. Seed based - correlation coefficient changes
  2. ASL - % change
  3. MRS - % change
Time Frame: Twice per session in MRI Phase (pre-TMS and immediately post-TMS)
Population: as for outcome 1
Arm/Group | Low Frequency rTMS - Behavioral Phase | High Frequency rTMS - Behavioral Phase | High Frequency rTMS - MRI Phase
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) monitoring took place from participant consent to 3 weeks after final TMS session. The actual timeframe varied based on participant schedules and availability. Participants completed a TMS monitoring questionnaire before and after each TMS session, as well as 3 weeks after their final TMS session. Participants also completed a nursing assessment the morning of TMS appointments and had vitals taken at the end of each TMS appointment.
Description: AE collection was broken down by phase of the study (Behavioral vs. MRI), TMS Frequency (1Hz vs 10Hz), and Percentage of Motor Threshold (100%, 110%, Sham). Percentage of Motor Threshold (MT) corresponds with the milestones listed in the participant flow section.
Groups:
- Low Frequency rTMS - 100% MT - Behavioral Phase: Active 1Hz rTMS at 100% of motor threshold during the behavioral phase
- Low Frequency rTMS - 110% MT - Behavioral Phase: Active 1Hz rTMS at 110% of motor threshold during the behavioral phase
- Low Frequency rTMS - Sham - Behavioral Phase: Low Frequency rTMS, sham, during behavioral phase.
- High Frequency rTMS - 100% MT - Behavioral Phase: Active 10Hz rTMS at 100% of motor threshold during the behavioral phase
- High Frequency rTMS - 110% MT - Behavioral Phase: Active 10Hz rTMS at 110% of motor threshold during the behavioral phase
- High Frequency rTMS - Sham - Behavioral Phase: High Frequency rTMS, sham, during behavioral phase.
- High Frequency rTMS - 100% MT - MRI Phase: Active 10Hz rTMS at 100% of motor threshold during the MRI phase of the study.
- High Frequency rTMS - 110% MT - MRI Phase: Active 10Hz rTMS at 110% of motor threshold during the MRI phase of the study.
- High Frequency rTMS - Sham - MRI Phase: High Frequency rTMS, sham, during MRI phase.
Arm/Group | Low Frequency rTMS - 100% MT - Behavioral Phase | Low Frequency rTMS - 110% MT - Behavioral Phase | Low Frequency rTMS - Sham - Behavioral Phase | High Frequency rTMS - 100% MT - Behavioral Phase | High Frequency rTMS - 110% MT - Behavioral Phase | High Frequency rTMS - Sham - Behavioral Phase | High Frequency rTMS - 100% MT - MRI Phase | High Frequency rTMS - 110% MT - MRI Phase | High Frequency rTMS - Sham - MRI Phase
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/6 | 0/5 | 0/5 | 0/25 | 0/27 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/8 | 0/6 | 0/5 | 0/5 | 0/25 | 0/27 | 0/26
Other Adverse Events (participants affected / at risk) | 5/7 | 1/7 | 0/8 | 0/6 | 0/5 | 0/5 | 3/25 | 2/27 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Frequency rTMS - 100% MT - Behavioral Phase (N=7) | Low Frequency rTMS - 110% MT - Behavioral Phase (N=7) | Low Frequency rTMS - Sham - Behavioral Phase (N=8) | High Frequency rTMS - 100% MT - Behavioral Phase (N=6) | High Frequency rTMS - 110% MT - Behavioral Phase (N=5) | High Frequency rTMS - Sham - Behavioral Phase (N=5) | High Frequency rTMS - 100% MT - MRI Phase (N=25) | High Frequency rTMS - 110% MT - MRI Phase (N=27) | High Frequency rTMS - Sham - MRI Phase (N=26)
Headache (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Participants developed a headache during the rTMS session - stimulation was stopped upon request of participant. Expected, non-serious, related adverse event.
Headache and Dizziness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — Participant reported headache and dizziness. Expected, non-serious, related adverse event.
Hypomanic Episode (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant reported on 4/3/2017 that after orientation session on 3/13/17, she felt elevated mood and restlessness that lasted until the next day. Expected, non-serious, possibly related adverse event.
Involuntary Movement After TMS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participants showed involuntary motor activity (twitch in foot) after stimulation for motor threshold determination. Participants were withdrawn from the study and offered follow-up neurological assessment. Expected, non-serious, related AE.

LIMITATIONS AND CAVEATS:
Data collection closed 9/17/2019. Data have not yet been analyzed due to personnel turnover. There are currently no resources to complete data analysis. Data were transferred to a repository protocol for future analysis when resources are available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-30): https://cdn.clinicaltrials.gov/large-docs/92/NCT02231892/Prot_SAP_000.pdf